CLINICAL TRIAL: NCT01209013
Title: Multicenter, Prospective, Open-label, Single-arm Phase IIIb/IV Clinical Study on the Safety of Photodynamic Therapy With Porfimer Sodium for Injection for the Ablation of High-grade Dysplasia in Barrett's Esophagus
Brief Title: Safety of Photodynamic Therapy (PDT) in the Ablation of High-grade Dysplasia (HGD) in Barrett's Esophagus (BE)
Acronym: Oedisse
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor cancelled the study
Sponsor: Pinnacle Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-PO-PHOEST07-01
Record Dates: First submitted 2010-09-17; First posted 2010-09-24 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Barrett Esophagus
Keywords: PDT; porfimer sodium; BE
MeSH Terms: conditions — Barrett Esophagus | interventions — Endoscopy; Biopsy; X-Rays; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medlight PDT Balloon (Experimental)
  Interventions: Device: Medlight PDT Balloon; Procedure: Endoscopy; Procedure: Endoscopy with biopsy; Procedure: Electrocardiogram; Procedure: Chest x-ray; Procedure: Blood collection; Procedure: Tissue sample collection

INTERVENTIONS:
Device: Medlight PDT Balloon — Medlight PDT Balloon will be used once to apply the laser light treatment
Procedure: Endoscopy — Endoscopy will be performed to confirm eligibility, apply photodynamic therapy, assess esophageal condition and effectiveness of the therapy
Procedure: Endoscopy with biopsy — Endoscopy with collection of esophageal tissue will be performed at screening to confirm eligibility and at Week 13 (final visit) to assess effectiveness
Procedure: Electrocardiogram — Resting electrocardiogram will be performed at screening (unless one has been performed within 30 days prior to screening) to measure heart function
Procedure: Chest x-ray — A chest X-ray will be performed at screening (unless one has been performed within 90 days prior to screening) to provide several pictures of the chest to rule out any lung abnormalities
Procedure: Blood collection — Blood samples for laboratory tests will be taken to assess the overall condition
Procedure: Tissue sample collection — Esophageal tissue samples will be collected before the porfimer sodium injection and on four separate occasions after the injection (22-26 hour-, 40-50 hour-, 96-120 hour-intervals, and 13 weeks) to measure concentrations of oligomers in a subgroup of 12 patients.

SUMMARY:
Photodynamic therapy (PDT) uses a combination of a drug, porfimer sodium, and a light from a non heated laser. The activation of the drug is done by lighting of abnormal areas using a fiber optic device. The fiber optic device is a very fine fiber (like a fishing line) that permits transmission of light. The fiber optic device is inserted into a diffusing balloon device to ensure the good positioning of the fiber optic within the esophagus (food pipe). It is thought that the size and the flexibility of a new diffusing balloon device could improve the safety profile of the photodynamic treatment by reducing the risk of narrowing or closure of the food pipe (esophageal stenosis) sometimes occurring after treatment.

This research study will evaluate the safety and effectiveness of PDT with porfimer sodium using a new diffusing balloon device for light application in the removal of high-grade dysplasia (HGD, precancerous change in the food pipe tissue) in Barrett's esophagus (BE). This study will provide advanced knowledge about phototoxicity (reaction similar to sunburn) and esophageal stenosis, main risks with this therapy. It will involve 75 patients with HGD in BE across North America and Europe and will last between 13 and 16 weeks. In addition, concentrations of porfimer sodium in the esophageal tissue will be analyzed in a subgroup of patients.

DETAILED DESCRIPTION:
Patients with biopsy-confirmed HGD in BE will be evaluated to confirm eligibility. Prior to enrollment, all inclusion and exclusion criteria will be verified. Medical procedures including demographic information, medical/surgical history, concurrent medical conditions, physical exam (including vital signs, body weight, height, and skin color), degree of difficulty in swallowing; electrocardiogram, chest X-ray, clinical laboratory testing, concomitant medication intake and other therapy uses will be collected.

All patients will receive one course of PDT consisting of an intravenous injection of 2.0 mg/kg of porfimer sodium over 3-5 minutes followed by one or two endoscopic laser light applications. The first laser light application will be performed within 40-50 hours using a new diffusing balloon catheter. The second laser light application (without a diffusing balloon catheter) will be performed within 96-120 hours on those areas showing an insufficient response to the first application. Follow-ups (Weeks 4 and 13) will include some or all of the following procedures: physical exam; vital signs evaluation; body weight; endoscopy; skin, degree of difficulty in swallowing and esophageal stenosis assessment; and clinical laboratory check. All patients will be asked general open questions about any occurrence of adverse events, change in concurrent medical conditions, use of adjunctive therapy/procedure, and intake of concomitant medication. All patients will undergo rigorous systematic endoscopic biopsy surveillance at Week 13 (final visit).

Tissue concentration of oligomers (component of porfimer sodium) in normal and abnormal esophageal tissues will be determined in a subgroup of 12 patients. These patients will provide esophageal tissue samples before the porfimer sodium injection and on four separate occasions after the injection (22-26 hour-, 40-50 hour-, 96-120 hour-intervals, and 13 weeks).

All patients will be followed for three months.

ELIGIBILITY:
Inclusion Criteria:

* Patients are males or females aged 18 or older.
* Patients have been diagnosed with biopsy-proven HGD in BE.
* Non-menopausal or non-surgically sterilized female patients must have a negative serum beta-HCG at the time of entry into the study.
* Non-menopausal or non-surgically sterilized female patients must use a medically acceptable form of birth control.
* Patients must sign an Informed Consent Form, which must comply with the ICH guidelines and local requirements.

Exclusion Criteria:

* Patients who have previously received PDT for HGD in BE.
* Patients who have previously undergone radiation therapy to the chest.
* Patients with known porphyria or known hypersensitivity to porphyrins or any excipients of the porfimer sodium.
* Patients who have esophageal cancer or in whom esophageal cancer, lymph node involvement, or metastases cannot be ruled out based on the pathology report, endoscopic ultrasonography (EUS), computed tomography (CT) scan or other diagnostic methods used in current practice no more than 30 days prior to date of consent.
* Patients with any acute or chronic medical or psychological illnesses as judged clinically significant by the investigator to preclude PDT procedure.
* Patients with a presence or history of neoplasms (treated during the last five years prior to study entry) other than carcinoma in situ of the cervix or basal carcinoma of the skin.
* Patients with esophageal strictures, esophageal diverticula, esophageal or gastric varices.
* Patients with known contraindications to analgesia or endoscopy.
* Patients with blood parameters of Grade 3 or higher on the Common Terminology Criteria for Adverse Events (CTCAE).
* Patients with unstable cardiovascular disease (Class III and IV cardiovascular disease according to the New York Heart Association's functional criteria).
* Patients with esophageal ulcers > 1 cm in diameter.
* Patients with tracheoesophageal or bronchoesophageal fistula.
* Patients with chronic/acute dermatologic conditions (e.g., urticaria, eczema, sunburn).
* Patients under anticoagulant therapy (only for the subgroup of 12 patients who will consent to provide tissue samples in order to determine the concentrations of oligomers).
* Patients with severe renal or hepatic impairment with parameters of Grade 3 or higher on the CTCAE.
* Patients who have been treated with any investigational drug during 60 days prior to the screening visit.
* Patients who are unable or unwilling to complete the follow-up evaluations required for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Incidence of phototoxicity reaction | 3 months
Incidence of esophageal stenosis | 3 months

SECONDARY OUTCOMES:
Proportion of patients with complete ablation (removal) of high-grade dysplasia | 3 months
  Complete ablation of high-grade dysplasia (pre-cancerous tissue) will be evaluated by biopsy
Proportion of patients with adverse events as a measure of safety | 3 months
Measure oligomer concentrations | 3 months